CLINICAL TRIAL: NCT01903980
Title: Epipericardial Fat Necrosis: A Misdiagnosed Condition
Acronym: epipericardial
Status: Completed | Type: Observational
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Karina de Souza Giassi, MD, Hospital Sirio-Libanes
Other Study IDs: Epipericardial Fat Necrosis; Pericardial Necrosis (Registry Identifier: Epipericardial Fat Necrosis)
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Epipericardial Fat Necrosis
Keywords: Epipericardial Fat Necrosis; Fat Necrosis; Chest Pain; Pericardial Necrosis; Pleuritic pain
MeSH Terms: conditions — Fat Necrosis; Chest Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EFN Cases: Cases of patients with epipericardial fat necrosis CT findings
  Interventions: Other: No intervention. It is a retrospective study

INTERVENTIONS:
Other: No intervention. It is a retrospective study — No intervention. It is a retrospective study

SUMMARY:
Epipericardial fat necrosis is a benign and self-limited condition that mainly curses with acute pleuritic chest pain and therefore must be an important differential diagnosis for patients in emergency department (ED). The knowledge of characteristics symptoms and correct management may avoid misdiagnosis or mistakes with other severe conditions like pulmonary embolism, pericarditis or acute coronary disease.

Despite the importance of this entity, only fewer than 40 cases have been reported since 1957, when the condition was first described.

We have seen a couple of similar cases in our institution during a short period of time, and we suspect that these numbers doesn't mean the real prevalence of epipericardial fat necrosis, so maybe this condition could be underdiagnosed. Instead, there isn't a study that tried to estimate an incidence of this entity.

ELIGIBILITY:
Inclusion Criteria:

* patients with imaging criteria of EFN (defined as a round fat attenuation lesion with peripheral stranding located in the epipericardial fat)

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the emergency department of SIrio-Libanes Hospital who performed a chest CT due to any reason
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determinate the incidence of epipericardial fat necrosis | 18 months

SECONDARY OUTCOMES:
Identify misdiagnosed cases of epipericardial fat necrosis | 18 months

OTHER OUTCOMES:
Describe Clinical and Radiological data of epipericardial fat necrosis | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital Sirio Libanes, São Paulo, São Paulo
  - Hospital Sirio-Libanes, São Paulo, São Paulo

REFERENCES:
- See also: Abstract of the initial research presented at 2013 ATS conference — http://www.atsjournals.org/doi/pdf/10.1164/ajrccm-conference.2013.187.1_MeetingAbstracts.A4913